CLINICAL TRIAL: NCT01342367
Title: A Feasibility Study of Oral Hormonal Therapy and Radiation for Non-metastatic, Intermediate or High Risk Prostate Cancer in Men 70 and Older or With Medical Comorbidities
Brief Title: Feasibility of Hormones and Radiation for Intermediate or High Risk Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-625-A
Record Dates: First submitted 2011-04-15; First posted 2011-04-27 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Dutasteride; Finasteride; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Androgen Therapy (Experimental): Subjects will receive two oral hormonal drugs (bicalutamide with dutasteride or bicalutamide with finasteride)
  Interventions: Drug: Bicalutamide; Drug: Dutasteride; Drug: Finasteride; Radiation: Radiation

INTERVENTIONS:
Drug: Bicalutamide — Bicalutamide 50 mg orally daily with either dutasteride or finasteride for 2 months. After two months of treatment bicalutamide with either dutasteride or finasteride will be taken along with radiation. After completion of radiation, bicalutamide will be stopped.
  Other Names: Casodex
Drug: Dutasteride — Dutasteride 0.5 mg orally will be taken daily with bicalutamide for 2 months. After two months of treatment dutasteride and bicalutamide will be taken along with radiation. After completion of radiation, dutasteride will be taken alone for two years.
  Other Names: Avodart; Jalyn
Drug: Finasteride — Finasteride 5 mg orally will be taken daily with bicalutamide for 2 months. After two months of treatment finasteride and bicalutamide will be taken along with radiation. After completion of radiation, finasteride will be taken alone for two years.
  Other Names: Propecia; Proscar
Radiation: Radiation — 7-8 weeks of radiation with bicalutamide and either dutasteride or finasteride.

SUMMARY:
The purpose of this study is see if quality of life is improved in patients receiving oral hormone therapy compared to standard of care. The study will also compare survival rates between patients receiving oral hormone therapy and those receiving standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 70 years and/or Charlson comorbidity index score > or = 2
* Pathologically (histologically) proven diagnosis of prostatic adenocarcinoma
* Two or more of the following intermediate risk features for recurrence, Gleason Score = 7, PSA 10-20 ng/ml, Clinical Stage T2b-T2c Percent positive biopsy cores > or = 50%
* One or more of the following high risk features for recurrence, Gleason Score 8-10, PSA > 20 ng/ml, Clinical Stage T3a-T4
* Clinically negative lymph nodes as established by imaging, nodal sampling, or dissection
* No evidence of bone metastases on bone scan
* History/physical examination via the Charlson Comorbidity Index within 60 days prior to registration
* Zubrod Performance Status 0-2
* Age > or = 18
* Baseline serum PSA within 60 days prior to registration
* Baseline serum testosterone obtained within 60 days prior to registration
* Study entry PSA and serum testosterone must not be obtained during the following time frames, 10-day period following prostate biopsy, following initiation of oral androgen manipulation, within 30 days after discontinuation of finasteride or dutasteride
* CBC/ differential obtained within 60 days prior to registration with adequate bone marrow function
* Patient must be able to provide study-specific informed consent prior to study entry
* Liver function parameters as follows, Total Bilirubin < or = 2 x institutional upper limit of normal, AST (SGOT) or ALT (SGPT) < or = 2 x institutional upper limit normal

Exclusion Criteria:

* Prior radical surgery (prostatectomy), high-intensity focused ultrasound (HIFU) or cryosurgery for prostate cancer
* Prior hormonal therapy, such as LHRH agonists (e.g., goserelin, leuprolide), antiandrogens (e.g., flutamide, bicalutamide), estrogens (e.g., DES), or bilateral orchiectomy
* Use of 5-alpha reductase inhibitors (finasteride, dutasteride) specifically prescribed for the treatment of prostate cancer
* Prior or concurrent cytotoxic chemotherapy for prostate cancer; prior chemotherapy for a different cancer is permitted
* Prior radiation, including brachytherapy, to the region of the prostate that would result in overlap of RT fields
* Active lupus or scleroderma
* Severe, active co-morbidity, including but not limited to,unstable angina within the last 6 months without subsequent corrective cardiovascular procedure,or acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Hepatic insufficiency with AST, ALT, or Bilirubin > 2 x upper limit of normal,clinical jaundice, and/or coagulation defects
* Acquired Immune Deficiency Syndrome (AIDS); note, however, that HIV testing is not required for entry into this protocol.Patients who are HIV seropositive but do not meet criteria for diagnosis of AIDS are eligible for study participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-12-17 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Liauw, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SOC Cohort: the standard of care GnRH agonist (SOC) included bicalutamide 50 mg daily with injectable LHRH agonist (e.g. leuprolide or goserelin). for total duration of 2 years and 4 months RT given 6-8 weeks
- Oral ADT Group: Combined androgen blockade in the oral ADT group was bicalutamide 50 mg daily with an oral 5-AR inhibitor (i.e. finasteride 5 mg, or dutasteride 0.5 mg daily), fo rtotal duration of 2 year sand 4 months RT given 6 8 weeks
Period: Overall Study
Arm/Group | SOC Cohort | Oral ADT Group
Started | 32 | 42
Completed | 30 | 40
Not Completed | 2 | 2
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- SOC Cohort: the standard of care GnRH agonist (SOC) included bicalutamide 50 mg daily with injectable LHRH agonist (e.g. leuprolide or goserelin). for total duration of 2 years and 4 months Bicalutamide given for 4 months RT given 6-8 weeks
- Oral ADT Group: Combined androgen blockade in the oral ADT group was bicalutamide 50 mg daily with an oral 5-AR inhibitor (i.e. finasteride 5 mg, or dutasteride 0.5 mg daily), fo rtotal duration of 2 year sand 4 months Bicalutamide given for 4 months RT given 6 8 weeks
- Total: Total of all reporting groups
Arm/Group | SOC Cohort | Oral ADT Group | Total
Number analyzed (Participants) | 30 | 40 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 40 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (1) | 72 (1) | 72 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 40 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 22 | 29 | 51
  White | 7 | 9 | 16
  Asian | 1 | 1 | 2
  Hispanic | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 40 | 70
Prostate-Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 17.9 [3 to 205] | 12.6 [4 to 48] | 15.3 [3 to 205]
Adult Comorbidity Evaluation [Count of Participants; unit: Participants] — The Adult Comorbidity Evaluation 27 (ACE-27) is a validated comorbidity instrument that provides a score (0-3; 1=mild, 2=moderate, 3=severe) based on the number and severity of medical comorbidities.
  Participants
    >=2 | 18 | 30 | 48
    <2 | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Was Measured by the Expanded Prostate Cancer Index Composite (EPIC) Hormonal Health-related Quality of Life Questionnaire
Description: Questionnaires were completed in writing by the patient. Questionnaires were administered at 1-2 months after initiation of hormonal treatment (before RT), at 3-4 months (during RT), and at 6 months after initiation of study therapy. Patients also completed questionnaires at 12, 18, and 24 months after completion of radiation therapy. Of primary interest were the baseline and 6 month and 24 month timepoints which are reported here.
  Scale scores could range from 0-100, with higher scores indicating better quality of life.
Time Frame: Baseline, 6 months, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOC Cohort | Oral ADT Group
Number analyzed (Participants) | 30 | 40
score on a scale
  Baseline | 92 (0.04) | 89 (0.04)
  6 month | 81 (0.07) | 88 (0.07)
  24 month | 83 (0.05) | 84 (0.05)

2. Secondary Outcome: Percentage of Participants Free From Biochemical Failure
Description: Increase in prostate-specific antigen (PSA) measured over time. Freedom from biochemical failure (FFBF) was defined from the time of enrollment until PSA failure occurs as defined by the Phoenix definition of a rise to 2 ng/mL above the nadir PSA value.
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | SOC Cohort | Oral ADT Group
Number analyzed (Participants) | 30 | 40
percentage of participants | 81 | 88

ADVERSE EVENTS:
Time Frame: from Baseline starting of Radiation, to 3 months post Rt, 6 months, 12 months and 24 months post Radiation, up to a total of 2 years and 4 months.
Arm/Group | SOC Cohort | Oral ADT Group
All-Cause Mortality (participants affected / at risk) | 8/30 | 7/40
Serious Adverse Events (participants affected / at risk) | 2/30 | 2/40
Other Adverse Events (participants affected / at risk) | 14/30 | 18/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC Cohort (N=30) | Oral ADT Group (N=40)
GI Toxicity (Gastrointestinal disorders) | 2 (2) | 2 (2) — GI bleeding and ulceration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC Cohort (N=30) | Oral ADT Group (N=40)
GI Toxicity (Gastrointestinal disorders) | 10 (10) | 12 (12) — Diarrhea, Abdominal pain
GU toxicity (Renal and urinary disorders) | 14 (14) | 18 (18) — Frequency, incontinence, urgency

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT01342367/Prot_SAP_000.pdf